CLINICAL TRIAL: NCT00000924
Title: A Phase II Randomized, Multicenter Protocol Evaluating Two Antiretroviral Regimens Containing Combinations of Protease Inhibitors, NRTIs, and an NNRTI
Brief Title: A Study to Compare Two Different Anti-HIV Drug Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 403; 11358 (Registry Identifier: DAIDS ES); P1001S (substudy); P1004S (substudy); PACTG 403
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Nevirapine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
This study compares 2 different anti-HIV drug regimens to determine which is the most effective in lowering the amount of HIV in the blood. The anti-HIV drugs used in this study are 2 protease inhibitors (nelfinavir and ritonavir), 2 nucleoside reverse transcriptase inhibitors (stavudine and didanosine), and 1 nonnucleoside reverse transcriptase inhibitor (nevirapine).

These drug combinations have been previously studied in adults, but there is limited information on how well they work in HIV-infected children. It is important to develop drug combinations which are effective at suppressing the HIV virus in children.

DETAILED DESCRIPTION:
The use of combination therapy with 2 or more antiretroviral agents has been strongly supported by recent studies in both children and adults. However, as of yet, few combinations of antiretrovirals have been studied in large cohorts of stable HIV-1 infected, antiretroviral-experienced children. Evidence suggests that viral suppression may be more difficult to achieve in children. Therefore, it is important to develop new drug combinations which can maximally suppress plasma HIV-1 RNA concentrations in children.

Patients are stratified by prior antiretroviral treatment (zidovudine [ZDV]/lamivudine [3TC] versus d4T/other treatment) and by age (under 24 months versus 24 months and older). Patients are then randomized to 1 of 4 treatment groups.

Arm A1: ddI/NFV/RTV (for prior ZDV/3TC-treated patients). Arm A2: ddI/NFV/RTV (for prior d4T/other-treated patients). Arm B1: d4T/NFV/NVP (for prior ZDV/3TC-treated patients). Arm B2: d4T/NFV/NVP (for prior d4T/other-treated patients). Treatment is administered for 48 weeks. At Weeks 2, 4, and then every 4 weeks thereafter, patients undergo physical examinations, and blood samples are drawn to measure viral load. [AS PER AMENDMENT 4/27/00: Patients in Arms A1 and A2 may continue to receive medication for an additional 24 weeks. While on the treatment extension, patients must continue their current schedule for study drug administration and completion of study visits. Patients in Arms A1 and A2 who have reached Week 44 participate in an enteric-coated ddI pharmacokinetic study as part of this 24-week extension. Patients who were enrolled in Arms A1 or A2 and who were taken off study after reaching Week 48 may be re-entered onto the study at Week 52 regardless of the number of weeks they have been off study.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are between 4 months and 21 years of age (consent of parent or guardian required if under 18).
* Are HIV-positive.
* Have a viral level of at least 4,000 copies/ml.
* Have a CD4 cell count of at least 750 (under 12 months of age), at least 500 (1 to 5 years of age), or at least 200 (6 years of age or older) cells/mm3 within the past 4 months or a CD4 percent of 15 percent or higher within the past 4 months.
* Have received the same continuous antiretroviral therapy for the past 16 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an active opportunistic and/or serious bacterial infection.
* Have been diagnosed with a malignancy.
* Have received prior treatment with certain antiretroviral medications.
* Are pregnant or breast-feeding.

Ages: 4 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wiznia, Study Chair
Locations (45):
- United States (42):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Earl K Long Early Intervention Clinic, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Result] King JR, Nachman S, Yogev R, Hodge J, Aldrovandi G, Hughes MD, Chen J, Wiznia A, Damle B, Acosta EP. Efficacy, tolerability and pharmacokinetics of two nelfinavir-based regimens in human immunodeficiency virus-infected children and adolescents: pediatric AIDS clinical trials group protocol 403. Pediatr Infect Dis J. 2005 Oct;24(10):880-5. doi: 10.1097/01.inf.0000180508.21918.8a. PMID 16220085